CLINICAL TRIAL: NCT02003131
Title: Safety and Feasibility Study of Mesenchymal Trophic Factor (MTF) for Treatment of Osteoarthritis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No enrollment
Sponsor: Translational Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBS-MTFOA-001
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; umbilical cord; mesenchymal; stem cells; trophic factors
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intra-articular knee injection of MTF (Other): Trophic factors from umbilical cord mesenchymal stem cells administered intra-articularly.
  Interventions: Biological: Trophic factors from umbilical cord mesenchymal stem cells
- Subcutaneous injection of MTF (Other): Trophic factors from umbilical cord mesenchymal stem cells administered subcutaneously once per week for 12 weeks.
  Interventions: Biological: Trophic factors from umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: Trophic factors from umbilical cord mesenchymal stem cells

SUMMARY:
Allogeneic mesenchymal trophic factors (MTF) from human umbilical cord tissue-derived mesenchymal stem cells (UC-MSC) injected into the knee joints of 20 patients (group 1) or injected subcutaneously into 20 patients (group 2) is a safe and useful procedure for inducing joint function improvements in osteoarthritis (OA) patients with grade 2, 3, or 4 radiographic OA severity.

DETAILED DESCRIPTION:
The proposed study will assess primary safety and secondary efficacy endpoints of allogeneic UC-MSC-derived MTF administered to two arms osteoarthritis patients with grade 2, 3, or 4 radiographic OA severity (20 per arm). The first arm will receive an intra-articular injection of MTF into the knee joint under fluoroscopy. The second arm will receive 12 subcutaneous MTF injections, once per week.

For both arms, the primary objective of safety will be defined as freedom from treatment associated adverse events for the period of one year. The secondary objective of efficacy will include evaluation at baseline and at months 3 and 12 of efficacy endpoints of joint function improvement as assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and ability to understand the planned treatment.
* Subjects 18 years of age or older with idiopathic or secondary osteoarthritis of the knee with grade 2, 3, or 4 radiographic severity, as defined by the modified Kellgren-Lawrence classification

Exclusion Criteria:

* Pregnant women or cognitively impaired adults.
* Presence of large meniscal tears ("bucket handle" tears), as detected by clinical examination or by magnetic resonance imaging.
* Inflammatory or post infectious arthritis.
* More than 5 degrees of varus or valgus deformity.
* Kellgren Lawrence grade 4 osteoarthritis in two compartments (the medial or lateral compartments of the tibiofemoral joint or the patellofemoral compartment) in persons over 60 years of age.
* Intra-articular corticosteroid injection within the previous 3 months.
* A major neurologic deficit.
* Serious medical illness with a life expectancy of less than 1 year.
* Prior admission for substance abuse
* Body Mass Index (BMI) of 40 kg/m2 or greater
* Patient receiving experimental medication or participating in another clinical study within 30 days of signing the informed consent
* In the opinion of the investigator or the sponsor the patient is unsuitable for cellular therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 12 months

SECONDARY OUTCOMES:
Number of participants with a change in joint function from baseline WOMAC assessment at 12 months | 12 months
Number of participants with a change in radiogrpahic evidence of knee OA from baseline Kellegren-Lawrence grading system at 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Paz-Rodriguez, MD, Principal Investigator — Translational Biosciences / Stem Cell Institute
Locations (1):
- Stem Cell Institute, Panama City, Panama